CLINICAL TRIAL: NCT06938620
Title: Efficacy of Flow Restrictors in Limiting Access of Liquid Medicines by Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Grady Health System (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CDC-NCEZID-6162
Record Dates: First submitted 2013-04-18; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Enhanced Child-safety Packaging
Keywords: Child Injury; Child-resistant Packaging; Pediatric Poisoning; Medication Safety; Injury Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bottle with a flow restrictor (Experimental): Bottle with 1 of 3 randomly assigned flow restrictor designs (FR-bottle)
  Interventions: Other: Bottle with a flow restrictor
- Control bottle (Active Comparator): Traditional bottle either no cap or an incompletely-closed child-resistant cap
  Interventions: Other: Control bottle

INTERVENTIONS:
Other: Bottle with a flow restrictor — Flow restrictors added to liquid medicine bottles to determine whether they limit accessibility of liquid bottle contents to young children compared with control bottles without flow restrictors.
  Arms: Bottle with a flow restrictor
Other: Control bottle — Traditional bottle either no cap or an incompletely-closed child-resistant cap
  Arms: Control bottle

SUMMARY:
This study aimed to assess whether adding flow restrictors, adapters added to the neck of a bottle to limit the release of liquid, affects the proportion of preschool-aged children who can access liquid bottle contents, the amount accessed, and the time required for children to empty the bottles compared with traditional bottles without flow restrictors.

DETAILED DESCRIPTION:
Unsupervised ingestion of medications by young children is an important public health concern, leading to tens of thousands of emergency department visits and many more calls to poison control centers each year. Current knowledge on the specific circumstances in which young children gain access to medications is limited; however, a number of studies have shown that improper replacement of child-resistant packaging (CRP) by a caregiver leads to a substantial number of these incidents. Beginning in 2011, several pharmaceutical manufacturers introduced flow restrictors on over-the-counter (OTC) infants' acetaminophen; however, the efficacy of flow restrictors in limiting accessibility of liquid medicines by young children has not been formally assessed.

This study sought to determine whether adding flow restrictors, adapters added to the neck of a bottle to limit the release of liquid, to liquid medicine bottles can provide additional protection against unsupervised medicine ingestions by young children. A modified version of the standard child test protocol for re-closeable packages outlined in the Poison Prevention Packaging Act (PPPA protocol) was used to assess the efficacy of flow restrictors in limiting children's access to liquid medicines. Preschool-aged children participated in two 10-minute trials in which they were asked to try to "get everything out" of bottles filled with test liquid (a food product with similar flow characteristics to liquid medicine). Randomized block design was used to assign specific bottles to participants. Each child tested an uncapped bottle with a flow restrictor (FR-bottle) for one trial (1 of 3 designs randomly assigned). For the other trial, the child tested a control bottle (a traditional bottle either no cap or an incompletely-closed child-resistant cap). The amount of liquid the child removed from each bottle was measured and the time required to empty bottles was recorded. If flow restrictors limit the amount of liquid a young child can access, even when the outer child-resistant cap is not fully secured, their use could potentially be expanded to other liquid medicines.

ELIGIBILITY:
Inclusion Criteria:

* Attends one of the participating preschools
* Is between 36 - 59 months of age
* Is an English speaker

Exclusion Criteria:

* Has an obvious or overt, temporary or permanent, injury, illness, or physical or mental disability
* Has known allergies/restrictions to ingesting any ingredients in the test liquid

Ages: 36 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Proportion of children who removed specified amounts of test liquid from FR-bottles compared with control bottles | 0 days
  Proportion of children who emptied bottles, removed ≥ 25 mL, and who removed ≥ 5 mL of liquid from FR-bottles compared with control bottles

SECONDARY OUTCOMES:
Time required to empty the bottles | 0 days
  Proportion of children who emptied bottles, removed ≥ 25 mL, and who removed ≥ 5 mL of liquid from FR-bottles compared with control bottles
Proportion of liquid removed from bottles | 0 days
  Proportion of children who emptied bottles, removed ≥ 25 mL, and who removed ≥ 5 mL of liquid from FR-bottles compared with control bottles
Approaches used to remove liquid from bottles | 0 days
  Proportion of children who emptied bottles, removed ≥ 25 mL, and who removed ≥ 5 mL of liquid from FR-bottles compared with control bottles
Differences in proportions of children who removed specified amounts of liquid by age, sex, and site | 0 days
  Proportion of children who emptied bottles, removed ≥ 25 mL, and who removed ≥ 5 mL of liquid from FR-bottles compared with control bottles

OTHER OUTCOMES:
Amount of test liquid removed from individual FR-bottle designs | 0 days
  Proportion of children who emptied bottles, removed ≥ 25 mL, and who removed ≥ 5 mL of liquid from FR-bottles compared with control bottles

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Budnitz, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention